CLINICAL TRIAL: NCT04738513
Title: One Year Clinical Evaluation of New Gradient Technology Monolithic Zirconia (5Y-TZP/3Y-TZP) Crowns in Dental Esthetic Zone With Vertical Versus Conventional Preparation Techniques (Randomized Clinical Trial)
Brief Title: One Year Clinical Evaluation of New Gradient Technology Monolithic Zirconia (5Y-TZP/3Y-TZP) Crowns in Dental Esthetic Zone With Vertical Versus Conventional Preparation Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatalla Ahmed Emad ElGendy, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 351020
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Single Anterior Crowns; Badly Decayed Teeth; Endodontically Treated Teeth; Spacing Between Anterior Teeth; Malposed Teeth(Tilted,Overerupted,Totated,Etc.)
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional preparation technique (Active Comparator): Monolithic Zirconia (5Y-TZP/3Y-TZP) Crowns using conventional preparation technique.
  Interventions: Procedure: Conventional Preparation technique
- Vertical preprartion (Experimental): Monolithic Zirconia (5Y-TZP/3Y-TZP) Crowns using Vertical preparation technique.
  Interventions: Procedure: Vertical preparation technique

INTERVENTIONS:
Procedure: Vertical preparation technique — Teeth in dental esthetic zone will receive Monolithic Zirconia (5Y-TZP/3Y-TZP) Crowns using vertical preparation technique.
  Other Names: Vertiprep
  Arms: Vertical preprartion
Procedure: Conventional Preparation technique — Teeth in dental esthetic zone will receive Monolithic Zirconia (5Y-TZP/3Y-TZP) Crowns using conventional preparation technique.
  Arms: Conventional preparation technique

SUMMARY:
The aim of this study is to evaluate the clinical behavior of zirconia crowns in dental esthetic zone with vertical versus conventional preparation techniques using a new gradient technology monolithic zirconia (5Y-TZP/3Y-TZP).

DETAILED DESCRIPTION:
Introduction: A good relationship between dental restorations and the periodontium is one of the most important aspects to ensure clinical success both in terms of esthetics and function. Dental preparation for fixed prostheses can take various forms classified as horizontal preparation with a defined margin (chamfer), or vertical, or without a margin/finish line. According to some clinical reports, vertical preparation technique provides an increases in the gingival thickness and a greater stability of the gingival margin. Moreover, vertical preparation is characterized by being more conservative with tooth structure. Also, taking impressions is easier since it is a finish area and not a defined line.

Null hypothesis:

1. There will be no difference between vertical and conventional preparations in the clinical behavior of zirconia crowns in dental esthetic zone at baseline,3,6,9,12 months evaluation.
2. There will be no difference between vertical and conventional preparations in the patient satisfaction of zirconia crowns in dental esthetic zone at baseline,3,6,9,12 months evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. From 21-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations.
3. Psychologically and physically able to withstand conventional dental procedures.
4. Patients with teeth problems indicated for all ceramic crowns in esthetic zone;

   1. Badly decayed teeth
   2. Teeth restored with large filling restorations
   3. Endodontically treated teeth
   4. Malformed teeth
   5. Malposed teeth (Tilted, over-erupted, rotated, etc.)
5. Able to return for follow-up examinations and evaluation.
6. Thick gingival biotype.

Exclusion Criteria:

1. Patient less than 21or more than 50 years.
2. Patient with active resistant periodontal diseases.
3. Patients with poor oral hygiene and uncooperative patients.
4. Pregnant women.
5. Patients in the growth stage with partially erupted teeth.
6. Psychiatric problems or unrealistic expectations.
7. Patient with periodontal problems.
8. Patients with malocclusion or parafunctional habits.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Marginal integrity | 1 year
  Measured by using Modified United States Public Health Service criteria (USPHS criteria)
  * Alpha (A) the explorer does not catch when drawn across the surface of the restoration toward the tooth, or, if the explorer does not catch, there is no visible crevice along the periphery of the restoration (visual inspection explorer)
  * Bravo (B) the explorer catches and the is visible evidence of the crevice, which the explorer penetrates, indicating that the edge of the restoration does not adapt closely to the tooth structure. The dentin and/or the base is not exposed, and the restoration is not mobile ( visual inspection and explorer)
  * Charlie (C) the explorer penetrates crevice defect extended to the dento-enamel junction (explorer)

SECONDARY OUTCOMES:
Gingival discoloration | 1 year
  Measured by using Modified United States Public Health Service criteria (USPHS criteria)
  * Alpha (A) None,
  * Bravo (B) Slight discoloration, removable by finishing,
  * Charlie (C) Discoloration, localized not removable,
  * Delta (D) Strong discoloration in major parts of the margin not removable
Gingival inflammation | 1 year
  Measured by using Modified United States Public Health Service criteria (USPHS criteria) Alpha (A) Non, Bravo (B) Slight, Charlie (C) Moderate, Delta (D) Severe
Restoration color stability | 1 year
  Measured by using Modified United States Public Health Service criteria (USPHS criteria) Alpha(A) No change, Bravo(B) change in comparison to baseline condition
Secondary caries | 1 year
  Measured by using Modified United States Public Health Service criteria (USPHS criteria) Alpha (A) Non, Bravo (B) Caries present
patient satisfaction | 1 year
  Measured by Visual Analog Scale VAS (Questionnaire) a numerical scale from ("0" unsatisfied to "10" satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided